CLINICAL TRIAL: NCT05935696
Title: A Prospective Observational Study on the Role of Transthoracic Ultrasound in Differentiating Tuberculous From Malignant Pleural Effusion
Acronym: TUS-TBE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sarawak General Hospital (Other)
Collaborators: Hospital Queen Elizabeth, Kota Kinabalu, Sabah (Unknown); Institute of Respiratory Medicine Malaysia, Kuala Lumpur (Unknown); Hospital Serdang, Selangor (Unknown); University of Malaya (Other); Hospital Melaka, Melaka (Unknown)
Responsible Party: Principal Investigator, Kho Sze Shyang, Dr., Sarawak General Hospital
Other Study IDs: TUS-TBE v4.0
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Pleural Effusion; Tuberculosis, Pleural; Malignant Pleural Effusion
Keywords: pleural effusion; transthoracic ultrasound; tuberculous pleural effusion
MeSH Terms: conditions — Pleural Effusion; Tuberculosis, Pleural; Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tuberculous Pleural Effusion: Tuberculous pleural effusion (TBE)
  if any of the following criteria is presence:
  * Histological evidence of caseating granuloma from pleural biopsy
  * Microbiological evidence (positive growth of Mycobacterium tuberculosis culture, positive TB-PCR, positive Xpert MTB/RIF) from pleural fluid or pleural biopsy specimen
  * In patients with positive sputum smear for acid fast bacilli, sputum positive for mycobacterium tuberculosis culture, sputum positive for Xpert MTB/RIF or TB-PCR with no apparent cause of an exudative pleural effusion
  Patient without histological or microbiological evidence who demonstrated therapeutic response to anti-tuberculosis drugs will not be accepted as TBE in current study.
- Malignant Pleural Effusion (Control): Malignant pleural effusion (MPE)
  if any of the following criteria is presence:
  • Histological or cytological evidence of specific histopathological diagnosis of malignancy from pleural biopsy Patient without histological or cytological evidence or malignancy (para-malignant) will not be considered as MPE in the context of this study.

SUMMARY:
Primary Endpoint

* To assess the prevalence and diagnostic performance of pre-determined echographic features in predicting the diagnosis of TBE from MPE.
* To determine the clinical, pleural fluid and echographic parameters that were different among TBE and MPE and to establish a clinical prediction model for TBE.

Secondary Endpoint

* To assess the correlation between pleural fluid parameters with ultrasound and medical thoracoscopic finding.
* To assess the optimal Pf ADA cut-off value to differentiate TBE from MPE in our region.

DETAILED DESCRIPTION:
Tuberculous (TBE) and malignant pleural effusion (MPE) is the commonest cause of exudative pleural effusion in Malaysia. Early differentiation between these two diagnoses is essential as TBE only requires drainage if symptomatic, whereas MPE would require tissue biopsy for diagnosis confirmation and molecular profiling. However, both TBE and MPE present almost similarly with lymphocytic exudates. Pleural fluid (Pf) indices such as adenosine deaminase (ADA) may allow differentiation between these two entities in appropriate clinical circumstances. However, Pf ADA may not readily be accessible in resource-limited regions and the optimal cut-off varies depending on the local prevalence of tuberculosis. As a result, TBE diagnosis in our region is still heavily dependent on the analysis of pre-existing clinical demographic data and Pf parameters, where ultimately requiring pleural biopsy for a confident clinical diagnosis.

Point-of-care predictors for TBE, such as ultrasound imaging appearance, may be helpful, but have rarely been described. Previous studies have demonstrated that a complex septated ultrasound pattern in lymphocytic pleural effusion is a potentially useful diagnostic predictor to differentiate TBE from MPE with a positive predictive value of 94% and likelihood ratio of 12.2 TBE diagnostic algorithms frequently include only clinical indices with Pf parameters such as Pf differential cell count, ADA, protein and lactate dehydrogenase (LDH). Incorporation of point-of-care ultrasound finding into the clinical diagnostic algorithm has not been extensively explored.

TBE is the result of a delayed type IV hypersensitivity reaction to mycobacterial protein; fibrin formation in the pleural cavity is largely driven by pro-inflammatory cytokines as well as a reduction of fibrinolytic activity due to pleural inflammation. In contrast, MPE is believed to be driven by a high degree of anaerobic metabolism leading to lactic acid production, rather than an inflammatory response. These different pathogenic mechanisms in TBE and MPE resulted in different pleural fluid parameters such as lower Pf glucose and pH with higher Pf LDH level in MPE when compared to TBE. We believed that this principle may be extrapolated to discriminative ultrasound findings between TBE and MPE.

The result from our retrospective pilot study found that the presence of echographic septation had an adjusted odds ratio of 9.28 in prediction of TBE diagnosis from MPE. Along with other clinical parameters (male gender, serum leucocyte counts 9 x 109/L or, pleural fluid protein 50g/L or more), these parameters collectively report a diagnostic accuracy of 79.61% (95% CI 74.13-84.38) for TBE. In a previous study conducted in region with low tuberculosis burden, pleural thickening of >1cm, pleural nodularity and diaphragmatic thickening of >7mm on transthoracic ultrasound were highly suggestive of MPE. However, not uncommonly, we observed similar pattern of pleural and diaphragmatic thickening in TBE patients in our region as well.

As TBE is a hypersensitivity process with significant inflammatory response, we hypothesize that echographic septation, in addition to pleural thickening and other sonographic findings, may be a good indicator, as part of a clinical prediction model to discriminate TBE from MPE in our region.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients 18 years old or more
* Undiagnosed exudative pleural effusion planning for diagnostic medical thoracoscopy

Exclusion Criteria:

* Patient less than 18 years old
* Patient for therapeutic medical thoracoscope (i.e., medical thoracoscopic adhesiolysis in patient with parapneumonic pleural effusion) in which diagnosis is already known.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients more than 18 years old who presented with undiagnosed pleural effusion scheduled for diagnostic medical thoracoscopy in all respective sites during first quarter of 2023 for six months will be considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Transthoracic ultrasound | 12 months
  To assess the prevalence and diagnostic performance of pre-determined echographic features in predicting the diagnosis of TBE from MPE.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarawak General Hospital, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No